CLINICAL TRIAL: NCT05588726
Title: Behavioral Intervention to Improve Insomnia Symptoms in Patients With Opioid Use Disorder
Brief Title: Improving Insomnia in Patients With Opioid Use Disorder
Acronym: OUDInsomnia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Staff no longer available to continue enrollment and other research activities
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 844147
Record Dates: First submitted 2022-10-13; First posted 2022-10-20 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Opioid Use Disorder; Insomnia
Keywords: Mindfulness
MeSH Terms: conditions — Opioid-Related Disorders; Sleep Initiation and Maintenance Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: This will be conducted as a parallel, single-blinded pilot study for reducing insomnia among patients with opioid use disorder who are stabilized on buprenorphine maintenance therapy. All subjects will participate in some form of insomnia treatment over a fourteen-day period (either the mindfulness relaxation therapy with sleep hygiene or only sleep hygiene for controls). Consent and screening will occur on Day -7, and the sleep diary will be assigned for baseline measurement. Randomization and survey baseline measurements from eligible participants will occur on Day -1, and participants will be randomized into one of two arms: one arm consisting of only the sleep hygiene intervention and the other consisting of both the sleep hygiene and mindfulness interventions. On Day 28, two weeks post-intervention(s), surveys will be emailed to participants to track any changes in sleep quality, mean buprenorphine dose, and frequency of non-prescribed opioid use.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Hygiene (Active Comparator)
  Interventions: Behavioral: Sleep Hygiene
- Mindfulness (Experimental)
  Interventions: Behavioral: Sleep Hygiene; Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Sleep Hygiene — Once weekly coaching calls with advice on sleep hygiene
Behavioral: Mindfulness — Once weekly coaching calls with advice on mindfulness
  Arms: Mindfulness

SUMMARY:
This randomized, 35-day research study (n=20) explores the effects of a simplified mindfulness intervention in opioid use disorder patients stabilized on buprenorphine maintenance therapy (BMT), aiming to alleviate insomnia, monitor BMT dose, and decrease non-prescribed opioid use. Patients tap along with their breathing at bedtime and practice sleep hygiene; controls do sleep hygiene only. Adherence will be monitored by a smartphone application.

DETAILED DESCRIPTION:
This research study is exploring the effects of a simplified mindfulness intervention in patients with opioid use disorder who are stabilized on buprenorphine maintenance therapy. This study aims to improve their sleep quality, monitor changes in buprenorphine dose, and decrease the frequency of non-prescribed opioids use. We will be enrolling a total of 20 patients who are above 18 years of age and have insomnia symptoms, opioid use disorder, and access to a smartphone. Patients will be asked to utilize a smartphone application which will allow us to monitor adherence; they will be asked to tap on the screen in time with their breathing before bedtime. Buprenorphine maintenance therapy is used to treat opioid use disorder (the buprenorphine will be prescribed by their healthcare provider as part of their standard clinical care and is not a research study intervention) by minimizing withdrawal symptoms, but symptoms of insomnia often persist. Symptoms of insomnia include difficulty falling/staying asleep, anxiety regarding sleep, or daytime sleepiness.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18
2. Diagnosed with Opioid Use Disorder
3. Stable on Buprenorphine Maintenance Therapy for at least 4 weeks
4. At least 3 nights of greater than 30 minutes of sleep onset latency
5. Speak English above 6th grade level
6. Access to smart device

Exclusion Criteria:

1. Inability to communicate verbally
2. Involved in another insomnia study
3. Medical or other factors that in the opinion of the study research team would interfere with their ability to participate in the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Sleep Onset Latency | Day 28
  Time to fall asleep as derived from the Sleep Diary

SECONDARY OUTCOMES:
Non-Prescribed Opioid Use | Days -1, 7, 14, and 28
  Non-Prescribed Opioid Use Questionnaire
Daytime Cravings | Days 1 through 14
  Smartphone app usage during the day

CONTACTS AND LOCATIONS:
Overall Officials: Nalaka Gooneratne, MD, MSc, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman School of Medicine, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ardame A, Bassaknejad S, Zargard Y, Rokni P, Sayyah M. Examine the Relationship between Mindfulness and Drug Craving in Addicts Undergoing Methadone Maintenance Treatment. Iran J Public Health. 2014 Mar;43(3):349-54. PMID 25988095
- [Background] Chakravorty S, Vandrey RG, He S, Stein MD. Sleep Management Among Patients with Substance Use Disorders. Med Clin North Am. 2018 Jul;102(4):733-743. doi: 10.1016/j.mcna.2018.02.012. PMID 29933826
- [Background] Dimsdale JE, Norman D, DeJardin D, Wallace MS. The effect of opioids on sleep architecture. J Clin Sleep Med. 2007 Feb 15;3(1):33-6. PMID 17557450
- [Background] Dunn KE, Finan PH, Andrew Tompkins D, Strain EC. Frequency and correlates of sleep disturbance in methadone and buprenorphine-maintained patients. Addict Behav. 2018 Jan;76:8-14. doi: 10.1016/j.addbeh.2017.07.016. Epub 2017 Jul 14. PMID 28735039
- [Background] Eacret D, Veasey SC, Blendy JA. Bidirectional Relationship between Opioids and Disrupted Sleep: Putative Mechanisms. Mol Pharmacol. 2020 Oct;98(4):445-453. doi: 10.1124/mol.119.119107. Epub 2020 Mar 20. PMID 32198209
- [Background] Garland EL, Hanley AW, Kline A, Cooperman NA. Mindfulness-Oriented Recovery Enhancement reduces opioid craving among individuals with opioid use disorder and chronic pain in medication assisted treatment: Ecological momentary assessments from a stage 1 randomized controlled trial. Drug Alcohol Depend. 2019 Oct 1;203:61-65. doi: 10.1016/j.drugalcdep.2019.07.007. Epub 2019 Aug 5. PMID 31404850
- [Background] Hallinan R, Elsayed M, Espinoza D, Veillard AS, Morley KC, Lintzeris N, Haber P. Insomnia and excessive daytime sleepiness in women and men receiving methadone and buprenorphine maintenance treatment. Subst Use Misuse. 2019;54(10):1589-1598. doi: 10.1080/10826084.2018.1552298. Epub 2019 May 26. PMID 31131668
- [Background] Kasasbeh E, Chi DS, Krishnaswamy G. Inflammatory aspects of sleep apnea and their cardiovascular consequences. South Med J. 2006 Jan;99(1):58-67; quiz 68-9, 81. doi: 10.1097/01.smj.0000197705.99639.50. PMID 16466124
- [Background] Khusid MA, Vythilingam M. The Emerging Role of Mindfulness Meditation as Effective Self-Management Strategy, Part 2: Clinical Implications for Chronic Pain, Substance Misuse, and Insomnia. Mil Med. 2016 Sep;181(9):969-75. doi: 10.7205/MILMED-D-14-00678. PMID 27612339
- [Background] Knutson KL, Ryden AM, Mander BA, Van Cauter E. Role of sleep duration and quality in the risk and severity of type 2 diabetes mellitus. Arch Intern Med. 2006 Sep 18;166(16):1768-74. doi: 10.1001/archinte.166.16.1768. PMID 16983057
- [Background] Kreek MJ, Reed B, Butelman ER. Current status of opioid addiction treatment and related preclinical research. Sci Adv. 2019 Oct 2;5(10):eaax9140. doi: 10.1126/sciadv.aax9140. eCollection 2019 Oct. PMID 31616793
- [Background] Lydon-Staley DM, Cleveland HH, Huhn AS, Cleveland MJ, Harris J, Stankoski D, Deneke E, Meyer RE, Bunce SC. Daily sleep quality affects drug craving, partially through indirect associations with positive affect, in patients in treatment for nonmedical use of prescription drugs. Addict Behav. 2017 Feb;65:275-282. doi: 10.1016/j.addbeh.2016.08.026. Epub 2016 Aug 15. PMID 27544697
- [Background] Serdarevic M, Osborne V, Striley CW, Cottler LB. The association between insomnia and prescription opioid use: results from a community sample in Northeast Florida. Sleep Health. 2017 Oct;3(5):368-372. doi: 10.1016/j.sleh.2017.07.007. Epub 2017 Aug 10. PMID 28923194
- [Background] Zimmerman M, McGlinchey JB, Young D, Chelminski I. Diagnosing major depressive disorder I: A psychometric evaluation of the DSM-IV symptom criteria. J Nerv Ment Dis. 2006 Mar;194(3):158-63. doi: 10.1097/01.nmd.0000202239.20315.16. PMID 16534432
- See also: SAMHSA Results from 2018 National Survey on Drug Use and Health — https://www.samhsa.gov/data/sites/default/files/cbhsq-reports/NSDUHNationalFindingsReport2018/NSDUHNationalFindingsReport2018.pdf